CLINICAL TRIAL: NCT05911880
Title: The Effect of a Plant-based Diet on the Active Rheumatoid Arthritis Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Fausto Sanchez Muñoz, Researcher in Medical Sciences D, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 211247
Record Dates: First submitted 2023-03-04; First posted 2023-06-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis; Diet, Healthy; Inflammatory Response
Keywords: vegetarian diet; cytokine; Arthritis; DAS-28; anti-inflammatory diet; pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Pain | interventions — Diet, Plant-Based; Diet, Mediterranean; Diet, Vegetarian; Diet, Vegan

STUDY DESIGN:
Intervention Model Description: Patients with established diagnosis of Rheumatoid Arthritis by the ACR 1987 or ACR/EULAR 2010 criteria, with mild to moderate disease activity measured by DAS-28 PCR (2.6-5.1), with personalized nutritional intervention, isocaloric and with modification of the percentage of proteins from plant origin (80%), for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjets with rheumatoid arthritis treated with a plant-based diet for 14 days (Experimental): The present study focuses on a dietary intervention in human subjects who have been diagnosed with rheumatoid arthritis for at least one year. The intervention consists of an individualized nutritional plan, isocaloric, and modifies the percentage of plant-based proteins to 80%, for 14 days, to evaluate if a plant-based diet affects the disease activity.
  The calorie intake given to each subject is calculated based on the average of 3 24-hour recalls and the basal energy expenditure using the Harris & Benedict formula. No medication modifications are made three months before and during the intervention.
  Fasting blood samples of blood are collected via venipuncture before and after the intervention to analyze the blood chemistry of six elements, a complete blood count, as well as to analyze the expression of microRNAs related to the disease and pro-inflammatory cytokines.
  In addition, body measurements (weight, body fat, visceral fat, and muscle) are taken using bioimpedance.
  Interventions: Behavioral: Plant-based diet for 14 days in patients with rheumatoid arthritis.

INTERVENTIONS:
Behavioral: Plant-based diet for 14 days in patients with rheumatoid arthritis. — Patients with low to moderate disease activity of rheumatoid arthritis (2.6-5.1 DAS28-CRP) underwent a dietary intervention consisting of an individualized, isocaloric, and plant-based diet with 57% carbohydrates, 25% lipids, and 18% proteins (80% of plant origin) for 14 days, without any modification of their medication regimen and with restricted consumption of processed foods.
  Other Names: Mediterranean diet; vegetarian diet; vegan diet; lacto-vegetarian diet; lacto-ovo-vegetarian diet

SUMMARY:
The increase in autoimmune diseases in Western countries has been linked to environmental factors, and diet is considered a modifier of rheumatoid arthritis (RA). A high-fat diet promotes systemic inflammation and alters the microbiome. Certain bacteria in the intestinal microbiota generate proinflammatory metabolites from components of red meat, eggs, and dairy products. However, fruits and vegetables can modulate the gut microbiota and have been associated with reduced inflammation in RA patients. The aim of this study is to determine the changes in RA activity associated with plant-based dietary modifications. The study will evaluate men and women aged 18 years and older with low, moderate, or severe RA activity, and the intervention will involve an individualized, isocaloric plant-based diet for 14 days. The 28-joint disease activity score index and c-reactive protein (DAS 28-PCR) will be used to determine disease severity, in addition to analyzing the expression of inflammatory cytokines and microRNAs associated with RA.

DETAILED DESCRIPTION:
The recent increase in autoimmune diseases in Western countries has seen environmental factors as important triggers of disease, as the genetic basis in affected populations has remained apparently constant. Diet has been seen as a modifying factor for several years in rheumatoid arthritis (RA).

A high-fat diet alters the structure of the microbiome even in the absence of obesity. However, it is also an important factor that promotes excessive accumulation of white adipose tissue (WAT) and systemic inflammation. For several decades, it has been evaluated how the intestinal microbiome participates in the metabolism of some components of the diet and has the potential to modify the circulating proinflammatory or anti-inflammatory mediators. In the context of patients with RA, it has been found that the bacterium Prevotella Copri, found in greater proportion in patients with newly diagnosed rheumatoid arthritis, generates a pro-inflammatory metabolite called N-trimethylamine oxide derived from choline and carnitine present in red meat, eggs, and dairy products. On the other hand, fruits and vegetables can modulate the gut microbiota through dietary fiber. The proportion of anti-inflammatory bacteria Faecalibacterium Prausnitzii, is higher in vegetarian diets, which has been seen in fecal flora as beneficial in patients with RA associated with reduced inflammation.

For several years, it has been reported in the literature that patients associate certain foods with increased or improved symptoms of the disease. However, a diet that combines several suggested strategies to reduce inflammation may represent a more significant intervention than just including specific foods in the diet. The role of the plant-based diet on RA activity has not been fully elucidated.

Based on this background, the objective of this work will be to determine the decrease in RA activity associated with plant-based dietary modifications. To carry out this protocol, women and men aged 18 and over with low, moderate, or severe rheumatoid arthritis activity will be evaluated. For dietary intervention, at the beginning of treatment, patients will be evaluated anthropometrically (weight, height, body mass index, waist and hip circumference, waist-hip index, percentage of total fat, visceral fat, and percentage of muscle), and a basal blood sample will be taken at the end of the procedure. The kilocalories typically consumed will be calculated through a 24-hour reminder to set your personalized meal plan. A dietary table will be made with the following distribution of macronutrients: carbohydrates 57%, protein 18%, and lipids 25%. Subsequently, the food will be distributed in an equivalent distribution table, complying with the kilocalories and the percentage of macronutrients established. The consumption of food of animal origin will be reduced, replacing this protein with vegetable protein.

The intervention will be carried out for 15 days, the menu will be modified at 7 days of intervention following the same specifications. At the end of the treatment, the patients will be evaluated under the same anthropometric conditions, and blood sampling for laboratory analyses. To determine the severity of the pathology, the DAS (Disease Activity Score) index will be used. A scale that measures RA activity. This scale influences the tumor and painful joint count on 28 joints, the rate of globular sedimentation (GSR), and the evaluation of the disease by the patient. This scale has a value of 0.0 to 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age.
* Established diagnosis of rheumatoid arthritis according to American College Rheumatoid (ACR) 1987 or ACR/European Alliance of Associations for Rheumatology (EULAR) 2010 criteria.
* Disease activity according to DAS 28 (defined as all > 2.6).

Exclusion Criteria:

* Systemic autoimmune superposition syndrome (with the exception of: fibromyalgia, thyroid pathology, Type 1 Diabetes Mellitus, syndrome Sjögren and antiphospholipid syndrome)
* Patients on treatment with coumarins
* Patients with cancer, chronic hepatitis, HIV, pregnancy
* Weight variations associated with diet in last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in disease activity by DAS28 at 14 days after with a plant-based diet | 14 days
  Is a scoring system to evaluate disease activity and treatment response in rheumatoid arthritis (RA).
  The scores are divided as follows:
  0-2.5: Remission 2.6-3.2: Low activity 3.3-5.1: Moderate activity >5.1: high activity This evaluates the joint count of 28 painful and inflamed joints in conjunction with the value of C-reactive protein (mg/L).

SECONDARY OUTCOMES:
Change from baseline in C-Reactive Protein (CRP) by automated photometry at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  < 5 mg/L = Low
  ≥ 5 mg/L = High
  CRP (C-reactive protein) is a measure used to assess the presence and amount of inflammation in the body. The liver produces CRP, and its levels in the blood increase in response to acute or chronic inflammation. It is considered a non-specific marker of inflammation, meaning that its elevated levels can indicate various inflammatory conditions, such as infections, autoimmune diseases, chronic inflammatory disorders, and tissue damage.
  CRP levels are evaluated by obtaining a fasting peripheral blood sample, with a minimum fasting period of 8 hours, using the venipuncture technique. The analysis is conducted using automated photometry.
Change from baseline in Erythrocyte Sedimentation Rate (ESR) by automated photometry at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  2-26.00 mm/hr = Normal
  ≥ 26 mm/hr = High
  Erythrocyte Sedimentation Rate (ESR) is a measure used to assess the presence of inflammation in the body. ESR is a non-specific indicator of inflammation and is based on the principle that red blood cells tend to clump together and settle more rapidly in the presence of inflammatory substances. It measures the distance that red blood cells descend in a test tube within one hour.
  ESR levels are evaluated by obtaining a fasting peripheral blood sample, with a minimum fasting period of 8 hours, using the venipuncture technique. The analysis is conducted using automated photometry.
Change from baseline in glucose by automated photometry at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  74-106 mg/dL = Normal
  ≥ 106 mg/dL = High
  Measures blood glucose levels. Glucose is a type of sugar that is the main source of energy for the human body. Measuring glucose in a clinical chemistry study provides important information about glucose metabolism and blood sugar control.
  Glucose levels are evaluated by obtaining a fasting peripheral blood sample, with a minimum fasting period of 8 hours, using the venipuncture technique. The analysis is conducted using automated photometry.
Change from baseline in Uric acid automated photometry at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  2.40-5.70 mg/dL = Normal
  ≥ 5.71 mg/dL = High The parameter of uric acid in the blood is a measurement used in clinical chemistry to assess the levels of uric acid present in the body. Uric acid is a waste product generated by the breakdown of purines, which are substances found in certain foods and also occur naturally in the body.
  Uric acid is transported through the bloodstream and is primarily eliminated through the kidneys in the form of urine. To evaluate uric acid levels, a fasting peripheral blood sample is obtained using the venipuncture technique, with a minimum fasting period of 8 hours. The analysis is conducted using automated photometry.
Change from baseline in total cholesterol concentration by automated photometry at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  0-200 mg/dL = Normal
  ≥ 201 mg/dL = High
  The parameter of total cholesterol in the blood is a measurement used in clinical chemistry studies to assess cholesterol levels in the body. Cholesterol is a lipid substance that is essential for the body's functioning, but elevated levels can increase the risk of cardiovascular diseases.
  Total blood cholesterol includes both HDL (high-density lipoprotein) cholesterol and LDL (low-density lipoprotein) cholesterol. Additionally, the measurement of total cholesterol may also include a fraction of triglycerides, which are another type of lipid.
  To evaluate total cholesterol, a fasting peripheral blood sample is obtained using the venipuncture technique, with a minimum fasting period of 8 hours. The analysis is conducted using automated photometry.
Change from baseline in Atherogenic index at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  1-4 = Normal
  ≥5 = High The atherogenic index is a parameter used in blood chemistry analysis to assess the risk of cardiovascular disease. This index provides information about the ratio between LDL (low-density lipoprotein) cholesterol and HDL (high-density lipoprotein) cholesterol in the blood.
  The index is calculated by dividing the LDL cholesterol by the HDL cholesterol. A high atherogenic index indicates an elevated ratio of LDL cholesterol to HDL cholesterol, which may indicate an increased risk of cardiovascular disease. Conversely, a lower index falls within the normal range and suggests a healthier cardiovascular profile.
Change from baseline in body weight by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  RESULT SCALE:
  Kilograms The body weight is measured using bioimpedance; a technique employed to assess body weight and gather additional information about an individual's body composition. During a bioimpedance measurement, a low-intensity electrical current is passed through the body, and the resistance encountered by body tissues is measured.
  Bioimpedance measurement of body weight is based on the principle that electrical current flows more easily through tissues with higher water content, such as muscles, while encountering greater resistance in tissues with lower water content, such as body fat.
Change from baseline in waist-to-hip index by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  Result scale:
  Female <0.80 = Low 0.81-0.85 = Moderate 0.86 = High
  Male:
  <0.95 = Low 0.96-1 = Moderate
  1 = High
  The waist-to-hip ratio is a measurement used to assess body fat distribution. To calculate the waist-to-hip ratio, you divide the waist circumference by the hip circumference.
  The waist-to-hip ratio serves as a general indicator of body fat distribution.
Change from baseline in body mass Index (BMI) by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  Result scale:
  Underweight: BMI < 18.5 kg/m2 Normal weight: BMI 18.5 - 24.9 kg/m2 Overweight: BMI 25 - 29.9 kg/m2 Class I obesity: BMI 30 - 34.9 kg/m2 Class II obesity: BMI 35 - 39.9 kg/m2 Class III obesity (morbid obesity): BMI ≥ 40 kg/m2
  The body mass index (BMI) is a measurement used to assess whether a person has a healthy weight in relation to their height. It is calculated by dividing a person's weight in kilograms by the square of their height in meters (BMI = weight / height²).
  BMI provides a general estimate of a person's amount of body fat and is used to assess the risk of developing certain weight-related diseases, such as obesity and heart disease.
Change from baseline in body fat percentage by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  Result scale:
  Sex Age Low Normal High Very High Female 20-39 < 21.0 21.0 - 32.9 33.0 - 38.9 >39 Female 40-59 < 23.0 23.0 - 33.9 34.0 - 39.9 >40 Female 60-79 < 24.0 24.0 - 35.9 36.0 - 41.9 >42 Male 20-39 < 8.0 8.0 - 19.9 20.0 - 24.9 >25 Male 40-59 < 11.0 11.0 - 21.9 22.0 - 27.9 >28 Male 60-79 < 13.0 13.0 - 24.9 25.0 - 29.9 >30 The body fat percentage is a measurement that indicates the proportion of fat in relation to the total weight of a person's body. It is a significant measure for assessing body composition.
  It is calculated using bioimpedance.
Change from baseline in visceral fat by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  Result scale:
  5-9 kilograms = Normal 10-14 kilograms = High
  15 kilograms = Very high
  This measurement assesses the amount of specific body fat that accumulates in the abdomen and surrounding vital organs. It is obtained through bioimpedance.
Change from baseline in skeletal muscle percentage by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  The skeletal muscle percentage is a measurement that reflects the proportion of skeletal muscle in relation to the total body weight of an individual. It is a significant indicator used to evaluate body composition.
  Result scale:
  Sex Age Low Normal High Very high Female 18-39 < 24.3 24.3 - 30.3 30.4 - 35.3 >35.4 Female 40-59 < 24.1 24.1 - 30.1 30.2 - 35.1 >35.2 Female 60-80 < 23.9 23.9 - 29.9 30.0 - 34.9 >35 Male 18-39 < 33.3 33.3 - 39.3 39.4 - 44.0 >44.1 Male 40-59 < 33.1 33.1 - 39.1 39.2 - 43.8 >43.9 Male 60-80 < 32.9 32.9 - 38.9 39.0 - 43.6 >43.7 This measurement is calculated using bioimpedance technique.
Change from baseline in metabolic age by bioelectric impedance analysis at 14 days after with a plant-based diet | 14 days
  Result scale:
  Measured in years. Body age is determined based on your basal metabolism. It takes into account factors such as weight, body fat percentage, and skeletal muscle percentage to calculate a reference value. This value helps determine whether your body age is higher or lower than your actual age.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Sanchez, PhD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez
Locations (1):
- Instituto Nacional de Cardiología "Ignacio Chávez", Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT05911880/Prot_000.pdf
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT05911880/ICF_001.pdf